CLINICAL TRIAL: NCT01383967
Title: Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of Multiple-Ascending Doses of LY2979165 in Healthy Subjects
Brief Title: A Study of LY2979165 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13846; I4S-EW-HHCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- LY2979165 Part A, Cohort 1 (Experimental): 20 mg LY2979165 administered orally, daily for 14 days
  Interventions: Drug: LY2979165
- LY2979165 Part A, Cohort 2 (Experimental): 60 mg LY2979165 administered orally, daily for 14 days
  Interventions: Drug: LY2979165
- LY2979165 Part A, Cohort 3 (Experimental): 100 mg LY2979165 administered, orally daily for 14 days
  Interventions: Drug: LY2979165
- LY2979165 Part A, Cohort 4 (Experimental): 150 mg LY2979165 administered orally, daily for 14 days
  Interventions: Drug: LY2979165
- LY2979165 Part B, Cohort 5 (Experimental): Dose to be determined by safety review of doses administered in Part A, administered, orally daily for 14 days
  Interventions: Drug: LY2979165
- Placebo (Placebo Comparator): Administered orally, daily for 14 days in a ratio of 3:1 in each Cohort of Part A
  Interventions: Drug: placebo
- LY2979165 Part A, Cohort 6 (Experimental): 250 mg LY2979165 administered orally, daily for 14 days
  Interventions: Drug: LY2979165
- LY2979165 Part A, Cohort 7 (Experimental): 400 mg LY2979165 administered orally, daily for 14 days
  Interventions: Drug: LY2979165

INTERVENTIONS:
Drug: LY2979165 — Administered orally
  Arms: LY2979165 Part A, Cohort 1; LY2979165 Part A, Cohort 2; LY2979165 Part A, Cohort 3; LY2979165 Part A, Cohort 4; LY2979165 Part A, Cohort 6; LY2979165 Part A, Cohort 7; LY2979165 Part B, Cohort 5
Drug: placebo — Administered orally
  Arms: Placebo

SUMMARY:
This is a two part study. Part A is a multiple-ascending dose study in up to 6 different groups of healthy subjects, with approximately 12 subjects in each of the groups. Part A will allow investigation of up to 6 different doses of LY2979165. The drug will be administered for a total of 14 days. Subjects will be resident in the clinical research unit (CRU) from Day -1 (the day before dosing) until Day 15.

Part B will investigate a dose of LY2979165 previously administered in Part A in up to 12 subjects. The drug will be administered for a total of 14 days. In addition to the same assessments as would have been completed in Part A, subjects in Part B will also have cerebrospinal fluid samples taken from the lower lumbar region of their spine.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination. Female subjects for Part B (if performed) are at the site's discretion.
* Male subjects: Agree to use a reliable method of birth control during the study
* Female subjects: Women not of child-bearing potential due to surgical sterilisation(hysterectomy or bilateral oophorectomy or tubal ligation) or postmenopausal as defined by age greater than or equal to 45 years, with an intact uterus, not taken hormones or oral contraceptives for > 1 year, and either: Spontaneous amenorrhoea of >12 months, or Spontaneous amenorrhoea of 6-12 months with a follicle-stimulating hormone (FSH) level of >40 mIU/mL
* Are between the body mass index (BMI) of 18.5 and 29.9 kg/m^2, inclusive
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* History of clinically significant adverse drug reactions or "drug allergy" to more than 3 different types of systemically administered medications (all penicillins and cephalosporins may be considered 1 type of medication for this purpose) or known allergies to LY2979165 or it's constituents
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2979165
* Have a Bazett's corrected QT (QTcB) interval value of >450 msec (males) or >470 msec (females) or any abnormality in the screening 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure (at least 5 minutes in supine position) as determined by the investigator
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, immunological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Show evidence of significant active neuropsychiatric disease
* Have increased risk of seizures as evidenced by a history of: greater than or equal to one (1) seizure (except childhood febrile seizure), history of electroencephalogram with epileptiform activity, history of stroke; surgery to the cerebral cortex; or head trauma with loss of consciousness
* Have a history of alcohol or drug abuse
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Intended use of over-the-counter medication within 7 days prior to dosing or during the study with the exception of vitamins and mineral supplements (not providing >100% of the recommended dietary allowance [RDA]), or occasional paracetamol or acetaminophen. If this situation arises, inclusion of an otherwise suitable subject may be at the discretion of the sponsor.
* Intended use of herbal supplements or prescription medications, other than stable doses of thyroid or estrogen hormone replacement, within 14 days prior to dosing or during the study. If this situation arises, inclusion of an otherwise suitable subject may be at the discretion of the sponsor.
* Have donated blood of more than 450 mL within the last 3 months
* Subjects who meet at least 1 of the following criteria (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits): a) subjects who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), b) subjects unwilling to stop alcohol consumption 48 hours prior to dosing until the completion of the 14-day dosing period, or c) subjects unwilling to limit alcohol intake to no more than 3 units per day at other times during the study.
* Cigarette consumption of more than 10 cigarettes per day or unable/unwilling to abide by CRU smoking restrictions during admissions
* Any other condition, which in the opinion of the investigator, would preclude participation in the study

Additional criteria for Part B:

* Abnormalities in lumbar spine previously known or determined by screening lumbar x-ray (if conducted).
* History of clinically significant back pain, back pathology and/or back injury (for example, degenerative disease, spinal deformity or spinal surgery) that may predispose to complications or technical difficulty with lumbar puncture
* Have evidence or history of significant active bleeding or coagulation disorder or have taken non-steroidal anti inflammatory drugs or other drugs that affect coagulation or platelet function within 14 days prior to lumbar catheter insertion
* Have an allergy to lidocaine (Xylocaine®) or its derivatives
* Have medical or surgical conditions in which lumbar puncture is contraindicated

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant effects | Baseline to study completion (estimate of 5 months, study ran for 11 months)

SECONDARY OUTCOMES:
Pharmacokinetics, area under the concentration curve (AUC): Part A | predose, up to 24 hours on day 1, predose and 4 hours on day 3, predose, up to 24 hours on day 7, predose day 8, predose and 4 hours on day 10, predose day 12 and 13 and predose,up to 48 hours on and after day 14
Pharmacokinetics, maximum concentration (Cmax): Part A | predose, up 24 hours on day 1, predose and 4 hours on day 3, predose, up to 24 hours on day 7, predose day 8, predose and 4 hours on day 10, predose day 12 and 13 and predose, up to 48 hours on and after day 14
Pharmacokinetics, area under the concentration curve (AUC): Part B | predose, up to 24 hours on day 1, predose and 4 hours on day 3, predose day 8, predose and 4 hours on day 10, predose day 12 and 13 and predose, up to 48 hours on and after day 14
Pharmacokinetics, maximum concentration (Cmax): Part B | predose, up to 24 hours on day 1, predose and 4 hours on day 3, predose day 8, predose and 4 hours on day 10, predose day 12 and 13 and predose, up to 48 hours on and after day 14
Pharmacokinetics; maximum concentration (Cmax) for Cerebrospinal Fluid (CSF): Part B | Pre dose (baseline) and 9 hours post dose
Pharmacodynamics; maximum concentration (Cmax) for CSF: Part B | Pre dose (baseline) and 9 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore